CLINICAL TRIAL: NCT05780099
Title: Prospective Observational Study to Characterize Patients Treated at Internal Medicine Clinics
Acronym: MED-Cli
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Rovere Querini Patrizia, Director, IRCCS San Raffaele
Other Study IDs: MED-Cli
Record Dates: First submitted 2023-02-21; First posted 2023-03-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Disease; Cardiovascular Diseases; Infectious Disease; Critical Illness; Immunological Disease; Pregnancy Disease; Metabolic Syndrome; Chronic Disease
MeSH Terms: conditions — Respiration Disorders; Cardiovascular Diseases; Communicable Diseases; Critical Illness; Immune System Diseases; Metabolic Syndrome; Chronic Disease | interventions — Inosine Monophosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: patients treated at internal medicine wards
  Interventions: Other: Inpatient or Outpatient visit

INTERVENTIONS:
Other: Inpatient or Outpatient visit — Patients will be seen and treated at the clinics like in the usual care

SUMMARY:
Patients referred to internal medicine wards are becoming increasingly complex and fragile. Despite deep knowledge of their specific disorders, steps are required to improve overall management of their acute and chronic conditions. The main objective of the study is to identify demographic, clinical, laboratory and radiological markers of disease severity and activity in patients with diseases treated at general medicine wards (respiratory disease, immune-mediated disease, sepsis, metabolic disease, rare disease, frailty, pregnancy pathology) in order to improve their diagnosis, monitoring and treatment processes.

DETAILED DESCRIPTION:
Among the most prevalent internal diseases worldwide are metabolic, respiratory and infectious diseases. Despite important progress in the field of these diseases, their frequent coexistence leads to a state of so-called fragility, now recognised as a genuine pathological condition, and entails the need to optimise their management in order to ensure faster and more effective diagnostic processes and targeted treatment procedures. On the other hand, those less frequent and less defined from both a pathogenetic and a management point of view include immune-mediated diseases, rare diseases, and internist disorders of pregnancy. Many times, diagnostic and therapeutic algorithms validated for specific diseases are arbitrarily applied to less common diseases based on the similarity of the clinical picture. For example, indices of inflammation such as C-reactive protein and erythrocyte sedimentation rate, traditionally used as markers of inflammatory response to infection, are commonly used as surrogate markers of disease activity in non-infectious immune-mediated diseases, despite the fact that there are no studies demonstrating their specific usefulness in patients suffering from them. This often leads to inappropriate care choices, as they are not based on sufficient degrees of evidence for those specific diseases. Studies focusing on specific disease categories are necessary to identify disease-specific markers and thus target therapy in an informed manner. Both the most prevalent and the least characterised pathologies require the integrated work of third-level centres, such as the San Raffaele Hospital, which have a large number of patient referrals and can therefore make a concrete contribution to the advancement of knowledge of these pathologies and their management and make their mark in the international scientific community. To this end, a prospective observational study is being conducted aimed at the detailed characterisation of patients suffering from these pathologies, in order to identify possible risk factors and markers of severity that can guide the development of new diagnostic and therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Receving treatment at internal medicine departments (inpatient, outopatient, day hospital) of San Raffaele Hospital
* at least one suspected or confirmed diagnosis among:

  1. immune mediated disorder
  2. respiratory disorder
  3. metabolic disorder
  4. sepsis
  5. rare disorder (according to Italian Ministry of Health list)
  6. pregnancy-related disorder
  7. frailty defined as: either ≥2 CIRS (Cumulative Illness Rating Scale) Severity Index 10 or ≤70% Karnofsky scale

Exclusion Criteria:

* refusal to participate
* enrolment in other intervantional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in outpatient, inpatient or day hospital setting of internal medicine units at San Raffaele Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2031-09-10 (Estimated); Study Completion 2032-09-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with severe disease | The following variables will be collected during patient enrollment
  Identify demographic, clinical, laboratory and radiological markers of disease severity and activity

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ospedale San Raffaele, Milan
  - San Raffaele Hospital, Milan

IPD SHARING:
Plan to Share IPD: Undecided